CLINICAL TRIAL: NCT04272424
Title: Changing the Innate Consensus About Mesh Fixation in Trans-abdominal Preperitoneal Laparoscopic Inguinal Hernioplasty in Adults: Short and Long Term Outcome. Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zagazig university 3
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): laparoscopic hernioplasty with no fixation
  Interventions: Procedure: laparoscopic mesh fixation
- group B (Active Comparator): laparoscopic hernioplasty with tacker fixation
  Interventions: Procedure: laparoscopic mesh fixation
- group C (Active Comparator): laparoscopic hernioplasty with histoacryl fixation
  Interventions: Procedure: laparoscopic mesh fixation

INTERVENTIONS:
Procedure: laparoscopic mesh fixation — laparoscopic mesh fixation by non fixation,tacker and histoacryl

SUMMARY:
Introduction: Inguinal hernioplasty is the standard treatment for inguinal hernia. Mesh fixation is used to keep mesh in place for which various mesh fixation techniques have been used in laparoscopic inguinal hernia repair, but their effectiveness has remained inconclusive.

Aim of the work: Randomized comparative study comparing early and late outcome of different method of mesh fixation.

Methods: In Zagazig University Hospitals, over the period from July 2016 to July 2018, patients with with oblique inguinal hernias undergoing Tans abdominal preperitoneal technique were randomized into 3 groups: Group A; mesh non fixation . Group B; tacker mesh fixation Group C: Cyanoacrylic tissue glues (Histoacryl) mesh fixation Clinical effects were assessed by the following variables: intraoperative data, postoperative outcome as regard recurrence rate, postoperative complications, analgesic consumption, operation time, hospital stay, and patient costs. Follow up was 18 months.

DETAILED DESCRIPTION:
Inguinal hernias are the commonest hernia met in clinical practice and accounts for 75% of abdominal hernia. Inguinal hernia repair is regarded as the standard treatment for adult symptomatic inguinal hernia following the international guideline for groin hernia management in which mesh is used to reinforce inguinal floor. Surgical mesh repair can be performed by open or laparoscopic techniques. Lichtenstein repair is commonly applied for open approach whereas trans-abdominal preperitoneal repair (TAPP) and totally extra peritoneal repair (TEP) are commonly used for laparoscopic approach.

During the repair of an inguinal hernia, sutures or tacks are generally used to secure the prosthetic mesh in place. In TAPP repairs the peritoneum is closed using sutures or tacks. These mesh ﬁxation or peritoneal closure techniques may contribute to postoperative chronic pain presumably due to nerve irritation or entrapment .

Several techniques for mesh fixations have been used including suture, glue or self-gripping mesh for open hernia repair (OHR); metallic tack, absorbable tack, glue, suture, self-gripping mesh or even non-fixation techniques for laparoscopic hernia repair (LHR). Up to date, there have been eight systematic reviews and meta-analyses (SRMAs) on OHR (ie, glue vs suture (n=5) and self-gripping mesh vs suture (n=3) and one network meta-analysis (NMA For LHR, comparisons were tack and glue (n=6).

fixation versus no fixation (n=3) .Although evidences were interesting, the overall results were inconclusive. In mesh-based repair, flat mesh is recommended over three-dimension mesh, while self-gripping mesh is another alternative mesh..

Intraoperative strategies to reduce pain include the non-ﬁxation of mesh or the use of non-mechanical methods of mesh ﬁxation other than tacking or suturing, which may be less traumatic to the local tissue and less likely to cause local nerve entrapment. These non-mechanical methods include self-ﬁxating meshes or glue. Similarly, closing the peritoneum with sutures may be less traumatic than the use of tacks, thus resulting in less postoperative pain .

Once positioned, meshes are designed to be integrated in local tissue by a fibrotic reaction that gradually incorporates them. Therefore, a good fixation is essential to secure the mesh in its correct position, while the integration process occurs. The introduction of synthetic meshes and their proper fixation has reduced recurrence rates to below 5%. As a consequence, the most frequent postoperative morbidities have become mesh migration, chronic pain, infection, and seroma .

Cyanoacrylic glues ensure high-degree and strong bonding to biologic tissues .When they get in contact with blood or water contained in the tissue, they form a very tight cover, binding to the surface within 5-6 s Overall, tacks provide excellent fixation strength, and they are also easy to apply. Nevertheless, their use is associated with significant morbidity. The penetration of the abdominal wall, in fact, may cause nerve and vessel entrapment. Also, tacks are themselves foreign bodies introduced in the abdomen, so they may cause inflammatory reactions. As a result, a significant number of patients suffer from pain and develop adhesion in the postoperative period. Moreover, cases of migration of titanium tacks have been described. At present, absorbable tacks are connected to lower inflammation rates, adhesion formation, and migration so the use of titanium tacks is no longer advisable

Aim of the work:

to determine whether there is any clinical or statistical difference in outcomes and morbidity when mesh is ﬁxed or not during laparoscopic TAPP inguinal hernia repair. We will also compare different methods of mesh ﬁxation (i.e.no fixation, tacks (non-absorbable and absorbable), and histoacryl) and techniques of peritoneal closure in TAPP repairs (tacks/sutures).

Patients & Methods:

Our study is a randomized controlled clinical trial. It was conducted on sixty adult male patients presenting with oblique inguinal hernia admitted in general surgery department, faculty of medicine Zagazig university from June 2016 to June 2018.

All the patients in this study were performed under the same surgical team after fulfilling the consent of the operation and after acceptance of the faculty of medicine Zagazig ethical committee.

The patients were randomly divided into three groups Group (A): includes twenty patients: no mesh fixation. Group (B): includes twenty patients: fixation of the mesh by tacker Group C: includes twenty patients: fixation of mesh by histoacryl.

Types of outcome measures Primary outcomes: Hernia recurrence (clinical or radiological at any time point), Chronic pain: pain persisting beyond three months postoperatively and persisting numbness: numbness in the groin or testicle persisting beyond three months postoperatively Secondary outcomes: Length of surgery (in minutes), Immediate postoperative pain (visual analogue scale (VAS)/ pain score),Vascular/visceral injury at operation,Haematoma/seroma development in postoperative period, Length of hospital stay (in days),Urinary retention in immediate postoperative period, Wound infection/mesh infection at any time point and Recovery time to normal activity (in days)

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 20 to 50
* Both sex
* An uncomplicated oblique inguinal hernia.
* Unilateral hernia

Exclusion Criteria:

* Patients younger than 20 or older than 50 year old
* Patients with complicated hernia
* Bilateral hernia
* Recurrent hernia
* Patients with previous lower abdominal surgery.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
pain following lap hernioplasty with different method of fixation | 1.5 years
  pain on visual analogue score

SECONDARY OUTCOMES:
recurrence of the disease following lap hernioplasty with different method of mesh fixation | 1.5 years
  recurrent hernia

CONTACTS AND LOCATIONS:
Overall Officials: tamer A. alnaimy, MD, Principal Investigator — Zagazig University

IPD SHARING:
Plan to Share IPD: No